CLINICAL TRIAL: NCT04774601
Title: The Role of Ultrasound Elastography in the Assessment of Chronic Liver Disease in Children
Brief Title: Elastography in Chronic Liver Disease in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Khalf Mohamed, Resident, Assiut University
Other Study IDs: Elastography in liver disease
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic liver disease is a significant health issue among children and it can result in fibrosis, cirrhosis and liver failure. Since the prognosis and monitoring of these diseases are different from each other,, Conventional ultrasonography is preferred for the investigation of chronic liver diseases in children, as it is non-invasive, cheap, feasible and available. Elastography, an ultrasonographic non-invasive procedure that measures tissue stiffness.

DETAILED DESCRIPTION:
Chronic liver disease is a significant health issue among children and it can result in fibrosis, cirrhosis and liver failure. Since the prognosis and monitoring of these diseases are different from each other, The term chronic liver disease (CLD) implies a long standing irreversible change in the hepatic structure that may end in complications like cirrhosis leading to premature death. While liver needle biopsy is still recognised to be the gold standard for the assessment of liver fibrosis in the diagnosis and follow-up of chronic liver diseases, researchers tend to study non-invasive methods in the determination of liver fibrosis, as liver needle biopsy is an invasive, painful and expensive procedure, which can cause possible sampling errors and potential complications , Conventional ultrasonography is preferred for the investigation of chronic liver diseases in children, as it is non-invasive, cheap, feasible and available. Elastography, an ultrasonographic non-invasive procedure that measures tissue stiffness.

Liver fibrosis is a result of chronic damage, and attacks and remissions throughout the course of the disease trigger the formation of fibrosis. Apart from being a direct indicator of liver damage, fibrosis has an important role in the development of hepatocyte dysfunction and portal hypertension. In a clinical aspect, knowing the state and progress of fibrosis is important in the assessment of treatment response for the severity and the prognosis of the disease. The degree of fibrosis in the liver is important in the determination of prognosis, and management of the process in chronic liver disease. Patients with fibrosis benefit from treatment in case of early diagnosis.

Ultrasound Elastography is a non-invasive method.

ELIGIBILITY:
Inclusion Criteria:

1 - all patients referred to the radiology department over the estimated period of the study. 2 - males and /or females from ( 0 to 18 years ) 3 - have clinical or laboratory or histopathological evidence of chronic liver disease 4 - had undergone liver biopsy.

Exclusion Criteria:

1. - Patients males and or females older than 18 years
2. - Patients who hadn't undergone liver biopsy previously
3. - Patients with acute liver disease
4. - Patients with human immune- deficiency virus (HIV) co infection.
5. - patients with pacemaker (PM) or implantable cardioverter defibrillator (ICD) devices.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients males and /or females from ( 0 to 18 years ) have clinical or laboratory or histopathological evidence of chronic liver disease und had undergone liver biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Comparison the results of ultrasound elastography in chronic liver disease in children with histopathlogical findings . | Baseline
  evaluate liver stiffness as a marker of severity and duration of the underlying chronic liver disease in children to achieve early diagnosis and benefit from treatment .

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Mostafa Thabet, Professor, Study Chair — Assiut University; Prof.Mohamed koriem, Assistant professor, Study Chair — Assiut University

REFERENCES:
- [Background] Sonmez S, Bosat M, Yurtseven N, Yurtseven E. The role of elastography in the assessment of chronic liver disease in children. Afr Health Sci. 2019 Sep;19(3):2806-2811. doi: 10.4314/ahs.v19i3.57. PMID 32127854